CLINICAL TRIAL: NCT01698957
Title: A Simple Technique to Modify Maternal Uterine Artery Perfusion.
Brief Title: Maternal Uterine Artery Doppler Study
Status: Completed | Type: Observational
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: UA Doppler 2012
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Maternal-Fetal Exchange
Keywords: Pregnant women; Uterine Artery Doppler Velocimetry
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UA Doppler Velocimetry: Any patient eligible for an Ultrasound greater than or equal to 18 weeks gestation without a fetal or uterine anomaly.
  Interventions: Other: Any patient eligible for an Ultrasound greater than or equal to 18 weeks gestation without a fetal or uterine anomaly.

INTERVENTIONS:
Other: Any patient eligible for an Ultrasound greater than or equal to 18 weeks gestation without a fetal or uterine anomaly. — bilateral Uterine artery Doppler readings pre- and during blood pressure measurement

SUMMARY:
The purpose of this study is to detect if adding resistance to maternal blood flow from the arm will help increase the blood flow through the uterine arteries to the placenta and the baby.

DETAILED DESCRIPTION:
In the setting of uteroplacental insufficiency, there is little that can be done to increase blood flow through the uterus and placenta. Historically, women with growth restricted fetuses or oligohydramnios have been placed on bed rest. Unfortunately, this treatment modality has met with only limited success. Cardiologists have long recognized the simple act of making a fist or otherwise occluding blood flow through a limb dramatically increases a person's peripheral vascular resistance. If maternal peripheral resistance can be increased, perhaps the increased differential between the maternal peripheral vascular resistance and that of the uteroplacental unit will increase flow through the uterus and placenta.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women greater than or equal to 18 years old
* Able to speak and read English
* Have a singleton pregnancy greater than or equal to 18 weeks gestation

Exclusion Criteria:

* Multiple gestation
* Less than 18 weeks gestation
* Uterine anomalies
* Fetal anomalies
* Preeclampsia
* Hypertension
* Inability to have BP cuff on left arm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women greater than or equal to 18 weeks gestation and 18 years old eligible for an ultrasound without fetal or uterine anomalies
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Uterine Artery Doppler | at time of routine ultrasound
  The purpose of this study is to detect if adding resistance to maternal blood flow from the arm will help increase the blood flow through the uterine arteries to the placenta and the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Strong, MD, Principal Investigator — Obstetrix Medical Group
Locations (2):
- United States (2):
  - Phoenix Perinatal Associates, Glendale, Arizona
  - Phoenix Perinatal Associates, Phoenix, Arizona